CLINICAL TRIAL: NCT04661631
Title: Lung Ultrasound in COVID-19 Infection Screening for Patients With Indication of Emergency Surgery
Brief Title: Surgery and Lung Ultrasound in COVID-19 Infection
Acronym: SOUNDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Sponsor
Other Study IDs: 1601
Record Dates: First submitted 2020-12-07; First posted 2020-12-10 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-05

CONDITIONS: Ultrasonography; Lung Diseases; Surgical Procedure; Covid19; Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: conditions — Lung Diseases; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Lung ultrasound during the screening process for SARS-CoV-2 infection in patients with an indication for urgent surgery.

SUMMARY:
The first case of COVID-19 was identified on December 19 and the world is actually experiencing a pandemic. The surgical procedure in patients with SARS-CoV-2 infection involves the exposure of other patients and the group of health workers who face the care of the patient. Thus, screening with lung ultrasound is an alternative to identify patients with an established or suspected infection that requires urgent surgery. Therefore, the aim of this study is to determinate the operational characteristics of lung ultrasound during the screening process for SARS-CoV-2 infection in patients with an indication for urgent surgery.

DETAILED DESCRIPTION:
Surgical intervention of a COVID-19 patient involves the exposure of other patients and the group of health workers who face the care of the patient, which generates additional stress and a subsequent catastrophic respiratory and cardiovascular decompensation.

Managing a patient who is going to undergo a surgical procedure as he was infected, makes health care workers and other patients aware from the risk of infection by reinforcing precautions measures. However, it implies the waste of personal protective elements, and a subsequent chance of consuming the limited stocks of those elements.

Li, Y, et al., described transmission of COVID-19 in a thoracic surgery department. They were infected from a single patient, and from three-generation transmission eight more patients and eleven health care workers. 3 out of 9 patients were infected and none of the health care workers died.

Lei et al reported a case series of 34 patients undergoing surgical treatment during the incubation period of COVID-19. They all developed symptoms. 44% of the patients presented dyspnea in the following days and a third presented ARDS. Seven patients (21%) died.

In both reports it is clear that the failure to identify patients as COVID-19 infected patients prevented them from being managed with the proper precautions and preventive measures, and that health care workers did not use adequate personal protective elements. On the other hand, the reported outcome in both series was worse than the outcome in COVID-19 patients who did not required surgical treatment. This corresponds to anecdotal reports of cases in which manifestations occurred after surgery and did not have a favorable clinical course.

In addition to this, an exponential growth of the infection by the COVID-19 virus in Colombia and the large amount of unidentified contaminants, justifies the implementation of a system that allows the identification of patients with COVID-19 infection, with the purpose of a correct surgical management, isolation, and protection of health care workers and other patients.

Screening with lung ultrasound is an alternative to identify patients with an established or suspected infection that requires urgent surgery. Its diagnostic efficacy has not been well studied in a systematic way in the scientific literature. Its use has just been described in patients with established COVID-19 pneumonia. Therefore, a research study is proposed to determine the operational characteristics of lung ultrasound during the screening process of patients who are going to be operated urgently.

ELIGIBILITY:
Inclusion Criteria:

* Indication for surgery for any reason
* Coming from the emergency room or hospitalized for less than 72 hours

Exclusion Criteria:

* Prisoner
* Chronic pulmonary disease
* Heart failure
* Kidney failure
* Referred from another hospital with invasive mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who enter the Fundación Valle del Lili who require emergency surgery for any reason
Sampling Method: Probability Sample
Enrollment: 451 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
The best cut-off point for lung ultrasound to discriminate suspected cases of active SARS-CoV-2 infection | 14 days
  To identify the best cut-off point from lung ultrasound that allows the discrimination of suspected cases of active SARS-CoV-2 infection in patients undergoing an emergency surgical procedure since May 2020 at Fundación Valle del Lili Hospital, Cali, Colombia.

SECONDARY OUTCOMES:
Prevalence of active SARS-CoV-2 infection | 14 days
  Identify the prevalence of active SARS-CoV-2 infection in the group of patients undergoing an emergency surgical procedure.
Operational characteristics of lung ultrasound | 14 days
  Calculate the operational characteristics of lung ultrasound for the diagnosis of SARS-CoV-2 infection in the studied group of patients.
Operational characteristics of each of suspicious lung ultrasound findings | 14 days
  Calculate the operational characteristics of each of suspicious lung ultrasound findings for the diagnosis of SARS-CoV-2 infection in the group of patients studied
Cut-off point resulting from the lung ultrasound score | 14 days
  Identify the cut-off point resulting from the lung ultrasound score that discriminates between patients with suspected active SARS-CoV-2 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto F. García, MDMSc, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundación Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No
The research information will be for the exclusive use of Fundación Valle del Lili

REFERENCES:
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Zhang S, Diao M, Yu W, Pei L, Lin Z, Chen D. Estimation of the reproductive number of novel coronavirus (COVID-19) and the probable outbreak size on the Diamond Princess cruise ship: A data-driven analysis. Int J Infect Dis. 2020 Apr;93:201-204. doi: 10.1016/j.ijid.2020.02.033. Epub 2020 Feb 22. PMID 32097725
- [Result] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Result] van Doremalen N, Bushmaker T, Morris DH, Holbrook MG, Gamble A, Williamson BN, Tamin A, Harcourt JL, Thornburg NJ, Gerber SI, Lloyd-Smith JO, de Wit E, Munster VJ. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med. 2020 Apr 16;382(16):1564-1567. doi: 10.1056/NEJMc2004973. Epub 2020 Mar 17. No abstract available. PMID 32182409
- [Result] Wang Y, Wang Y, Chen Y, Qin Q. Unique epidemiological and clinical features of the emerging 2019 novel coronavirus pneumonia (COVID-19) implicate special control measures. J Med Virol. 2020 Jun;92(6):568-576. doi: 10.1002/jmv.25748. Epub 2020 Mar 29. PMID 32134116
- [Result] Anelli F, Leoni G, Monaco R, Nume C, Rossi RC, Marinoni G, Spata G, De Giorgi D, Peccarisi L, Miani A, Burgio E, Gentile I, Colao A, Triassi M, Piscitelli P. Italian doctors call for protecting healthcare workers and boosting community surveillance during covid-19 outbreak. BMJ. 2020 Mar 26;368:m1254. doi: 10.1136/bmj.m1254. No abstract available. PMID 32217525
- [Result] The Lancet. COVID-19: protecting health-care workers. Lancet. 2020 Mar 21;395(10228):922. doi: 10.1016/S0140-6736(20)30644-9. No abstract available. PMID 32199474
- [Result] Kimball A, Hatfield KM, Arons M, James A, Taylor J, Spicer K, Bardossy AC, Oakley LP, Tanwar S, Chisty Z, Bell JM, Methner M, Harney J, Jacobs JR, Carlson CM, McLaughlin HP, Stone N, Clark S, Brostrom-Smith C, Page LC, Kay M, Lewis J, Russell D, Hiatt B, Gant J, Duchin JS, Clark TA, Honein MA, Reddy SC, Jernigan JA; Public Health - Seattle & King County; CDC COVID-19 Investigation Team. Asymptomatic and Presymptomatic SARS-CoV-2 Infections in Residents of a Long-Term Care Skilled Nursing Facility - King County, Washington, March 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 3;69(13):377-381. doi: 10.15585/mmwr.mm6913e1. PMID 32240128
- [Result] Tong ZD, Tang A, Li KF, Li P, Wang HL, Yi JP, Zhang YL, Yan JB. Potential Presymptomatic Transmission of SARS-CoV-2, Zhejiang Province, China, 2020. Emerg Infect Dis. 2020 May;26(5):1052-1054. doi: 10.3201/eid2605.200198. Epub 2020 May 17. PMID 32091386
- [Result] Li R, Pei S, Chen B, Song Y, Zhang T, Yang W, Shaman J. Substantial undocumented infection facilitates the rapid dissemination of novel coronavirus (SARS-CoV-2). Science. 2020 May 1;368(6490):489-493. doi: 10.1126/science.abb3221. Epub 2020 Mar 16. PMID 32179701
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Lauer SA, Grantz KH, Bi Q, Jones FK, Zheng Q, Meredith HR, Azman AS, Reich NG, Lessler J. The Incubation Period of Coronavirus Disease 2019 (COVID-19) From Publicly Reported Confirmed Cases: Estimation and Application. Ann Intern Med. 2020 May 5;172(9):577-582. doi: 10.7326/M20-0504. Epub 2020 Mar 10. PMID 32150748
- [Result] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Result] Li YK, Peng S, Li LQ, Wang Q, Ping W, Zhang N, Fu XN. Clinical and Transmission Characteristics of Covid-19 - A Retrospective Study of 25 Cases from a Single Thoracic Surgery Department. Curr Med Sci. 2020 Apr;40(2):295-300. doi: 10.1007/s11596-020-2176-2. Epub 2020 Mar 30. PMID 32232652
- [Result] Lei S, Jiang F, Su W, Chen C, Chen J, Mei W, Zhan LY, Jia Y, Zhang L, Liu D, Xia ZY, Xia Z. Clinical characteristics and outcomes of patients undergoing surgeries during the incubation period of COVID-19 infection. EClinicalMedicine. 2020 Apr 5;21:100331. doi: 10.1016/j.eclinm.2020.100331. eCollection 2020 Apr. PMID 32292899
- [Result] Wang W, Xu Y, Gao R, Lu R, Han K, Wu G, Tan W. Detection of SARS-CoV-2 in Different Types of Clinical Specimens. JAMA. 2020 May 12;323(18):1843-1844. doi: 10.1001/jama.2020.3786. PMID 32159775
- [Result] Cao Y, Liu X, Xiong L, Cai K. Imaging and clinical features of patients with 2019 novel coronavirus SARS-CoV-2: A systematic review and meta-analysis. J Med Virol. 2020 Sep;92(9):1449-1459. doi: 10.1002/jmv.25822. Epub 2020 Apr 10. PMID 32242947
- [Result] Ai T, Yang Z, Hou H, Zhan C, Chen C, Lv W, Tao Q, Sun Z, Xia L. Correlation of Chest CT and RT-PCR Testing for Coronavirus Disease 2019 (COVID-19) in China: A Report of 1014 Cases. Radiology. 2020 Aug;296(2):E32-E40. doi: 10.1148/radiol.2020200642. Epub 2020 Feb 26. PMID 32101510
- [Result] Bernheim A, Mei X, Huang M, Yang Y, Fayad ZA, Zhang N, Diao K, Lin B, Zhu X, Li K, Li S, Shan H, Jacobi A, Chung M. Chest CT Findings in Coronavirus Disease-19 (COVID-19): Relationship to Duration of Infection. Radiology. 2020 Jun;295(3):200463. doi: 10.1148/radiol.2020200463. Epub 2020 Feb 20. PMID 32077789
- [Result] Ding X, Xu J, Zhou J, Long Q. Chest CT findings of COVID-19 pneumonia by duration of symptoms. Eur J Radiol. 2020 Jun;127:109009. doi: 10.1016/j.ejrad.2020.109009. Epub 2020 Apr 18. PMID 32325282
- [Result] Zhao W, Zhong Z, Xie X, Yu Q, Liu J. Relation Between Chest CT Findings and Clinical Conditions of Coronavirus Disease (COVID-19) Pneumonia: A Multicenter Study. AJR Am J Roentgenol. 2020 May;214(5):1072-1077. doi: 10.2214/AJR.20.22976. Epub 2020 Mar 3. PMID 32125873
- [Result] Zhou Z, Guo D, Li C, Fang Z, Chen L, Yang R, Li X, Zeng W. Coronavirus disease 2019: initial chest CT findings. Eur Radiol. 2020 Aug;30(8):4398-4406. doi: 10.1007/s00330-020-06816-7. Epub 2020 Mar 24. PMID 32211963
- [Result] Huang Y, Cheng W, Zhao N, Qu H, Tian J. CT screening for early diagnosis of SARS-CoV-2 infection. Lancet Infect Dis. 2020 Sep;20(9):1010-1011. doi: 10.1016/S1473-3099(20)30241-3. Epub 2020 Mar 26. No abstract available. PMID 32222164
- [Result] Wong HYF, Lam HYS, Fong AH, Leung ST, Chin TW, Lo CSY, Lui MM, Lee JCY, Chiu KW, Chung TW, Lee EYP, Wan EYF, Hung IFN, Lam TPW, Kuo MD, Ng MY. Frequency and Distribution of Chest Radiographic Findings in Patients Positive for COVID-19. Radiology. 2020 Aug;296(2):E72-E78. doi: 10.1148/radiol.2020201160. Epub 2020 Mar 27. PMID 32216717
- [Result] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Result] Lichtenstein DA, Malbrain MLNG. Lung ultrasound in the critically ill (LUCI): A translational discipline. Anaesthesiol Intensive Ther. 2017;49(5):430-436. doi: 10.5603/AIT.a2017.0063. Epub 2017 Nov 18. PMID 29151003
- [Result] Testa A, Soldati G, Copetti R, Giannuzzi R, Portale G, Gentiloni-Silveri N. Early recognition of the 2009 pandemic influenza A (H1N1) pneumonia by chest ultrasound. Crit Care. 2012 Feb 17;16(1):R30. doi: 10.1186/cc11201. PMID 22340202
- [Result] Peng QY, Wang XT, Zhang LN; Chinese Critical Care Ultrasound Study Group (CCUSG). Findings of lung ultrasonography of novel corona virus pneumonia during the 2019-2020 epidemic. Intensive Care Med. 2020 May;46(5):849-850. doi: 10.1007/s00134-020-05996-6. Epub 2020 Mar 12. No abstract available. PMID 32166346
- [Result] Soldati G, Smargiassi A, Inchingolo R, Buonsenso D, Perrone T, Briganti DF, Perlini S, Torri E, Mariani A, Mossolani EE, Tursi F, Mento F, Demi L. Proposal for International Standardization of the Use of Lung Ultrasound for Patients With COVID-19: A Simple, Quantitative, Reproducible Method. J Ultrasound Med. 2020 Jul;39(7):1413-1419. doi: 10.1002/jum.15285. Epub 2020 Apr 13. PMID 32227492
- [Result] Vetrugno L, Bove T, Orso D, Barbariol F, Bassi F, Boero E, Ferrari G, Kong R. Our Italian experience using lung ultrasound for identification, grading and serial follow-up of severity of lung involvement for management of patients with COVID-19. Echocardiography. 2020 Apr;37(4):625-627. doi: 10.1111/echo.14664. Epub 2020 Apr 15. PMID 32239532
- [Result] Buderer NM. Statistical methodology: I. Incorporating the prevalence of disease into the sample size calculation for sensitivity and specificity. Acad Emerg Med. 1996 Sep;3(9):895-900. doi: 10.1111/j.1553-2712.1996.tb03538.x. PMID 8870764